CLINICAL TRIAL: NCT06923904
Title: Potassium Nitrate Gel and Diode Laser in the Treatment of Dentinal Hypersensitivity
Acronym: PotassiumNitra
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, University of Pavia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PotassiumNitrateLaser
Record Dates: First submitted 2025-03-14; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Dentistry; Desensitization
Keywords: desensitizing treatment; diode laser; oral hygiene; dental sensitivity
MeSH Terms: interventions — Therapeutics; Lasers, Semiconductor

STUDY DESIGN:
Intervention Model Description: This will be a randomized clinical trial (RCT) with a split-mouth design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with dental sensitivity (Experimental): With a split-mouth design the dental elements will be divided into the Trial group, treated with a 980 nm diode laser and desensitizing topical gel, and the Control group, treated only with the same gel.
  Interventions: Other: Trial group, treated with a 980 nm diode laser and desensitizing topical gel

INTERVENTIONS:
Other: Trial group, treated with a 980 nm diode laser and desensitizing topical gel — The study aims to evaluate the actual efficacy of diode lasers in laser desensitization by comparing the topical gel Emoform Actisens, containing 5% potassium nitrate, alone and in combination with a diode laser.

SUMMARY:
Our aim will be to evaluate the actual efficacy of diode lasers in laser desensitization by comparing the topical gel Emoform Actisens, containing 5% potassium nitrate, alone and in combination with a diode laser. Dental hypersensitivity (DH) will be assessed pre- (T0) and post-treatment (T1) and at 1 month (T2), 3 months (T3), and 6 months (T4).

DETAILED DESCRIPTION:
This will be a randomized clinical trial (RCT) with a split-mouth design, involving 12 subjects, with two parallel groups. The dental elements will be divided into the Trial group, treated with a 980 nm diode laser and desensitizing topical gel, and the Control group, treated only with the same gel. DH will be assessed using the Shiff Air Index (SAI) and Visual Analog Scale (VAS).

ELIGIBILITY:
The inclusion criteria will be as follows: (a) a good standard of home oral hygiene and (b) at least two teeth affected by DH.

The exclusion criteria will be: (a) individuals taking pain relievers; (b) individuals undergoing orthodontic treatment; (c) non-vital teeth; (d) teeth with restorative materials; and (e) pregnant or breastfeeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
degree of dentin hypersensitivity | From enrollment to 6 months after desensitizing procedure
  assessed using the Dentine Hypersensitivity Experience Questionnaire (DHEQ). The DHEQ is a validated self-report tool designed to assess the impact of dentine hy-persensitivity on a patient's daily life, including the intensity and frequency of symptoms as well as the emotional, social, and practical effects on daily activities such as eating, drinking, and oral hygiene practices. The DHEQ consists of 15 questions, with responses rated on a numerical scale from 1 ("strongly disagree") to 7 ("strongly agree"). The final score is calculated out of a total of 105 points, with higher scores indicating a greater im-pact of dentin sensitivity on daily life.

IPD SHARING:
Plan to Share IPD: No
Data will be publish as aggregate data with descriptive and inferential statistics